CLINICAL TRIAL: NCT02559284
Title: A Comparative, Multicenter and Randomized Study Evaluating the Safety and Efficacy of RESPIMER® Netiflow® Versus Saline Solutions During Nasal Irrigation Following Bilateral Ethmoidectomy in the Treatment of Nasal Polyposis.
Brief Title: RESPIMER® Netiflow® vs. Saline Solutions During Nasal Irrigation Following Bilateral Ethmoidectomy (Nasal Polyposis)
Acronym: NETIFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire de la Mer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P0013
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Polyp of Ethmoidal Sinus; Surgery
Keywords: Saline Solution, Isotonic / Administration & dosage; Therapeutic Irrigation / methods; Postoperative Care / methods; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - Experimental (Experimental): Treatment Arm: 100 patients using Respimer® NetiFlow® solution as standard treatment for healing of nasal surgery wounds following an endoscopic ethmoidectomy as a postoperative care after ethmoid sinus surgery
  Interventions: Other: A postoperative care after ethmoid sinus surgery
- B - Comparator (Active Comparator): Control Arm: 100 patients using saline solution (0.9% NaCl) as standard treatment for healing of nasal surgery wounds following an endoscopic ethmoidectomy as a postoperative care after ethmoid sinus surgery
  Interventions: Other: A postoperative care after ethmoid sinus surgery

INTERVENTIONS:
Other: A postoperative care after ethmoid sinus surgery — A comparison of two products used for nasal cavity cleansing, at the rate of 4 washes/day (240mL per wash), as local postoperative care following endoscopic sinus surgery. This surgery, known as an ethmoidectomy, aims to improve sinus ventilation, treat the chronically infected area, and remove polyps that cause nasal obstruction.
  Detailed information concerning the purpose of nasal irrigation, as well as how to use and clean the device, will be given to patients upon inclusion.
  The nasal washing procedure will be as follow:
  * Washing both nostrils using 180mL of solution distributed equally on each side to remove crusting and clotting
  * Gentle blowing of the nose
  * Rinsing both nostrils with the remaining 60mL of solution distributed equally on each side (no nose-blowing).

SUMMARY:
The main objective of this study is to compare the effects of RESPIMER® NetiFlow® solution and device versus saline solution (0.9% NaCl), the standard treatment, used with RESPIMER® NetiFlow® device, both used postoperative care, in the context of ethmoid sinus surgery, at 14 days post-surgery.

DETAILED DESCRIPTION:
This is a comparative study between two postoperative treatments following ethmoid sinus surgery. The purpose of this study is to compare the effect of RESPIMER® NetiFlow® solution on nasal tissue repair versus saline solution (0.9% NaCl), the standard treatment.

The type of surgery selected for this study is total endoscopic ethmoidectomy. This is a frequently used standard surgery that requires nasal cleansing for an average of 28 days. This process allows the regeneration of the nasal epithelial lining of the wound (areas of exposed bone), as well as the healing of swelling and scarring due to the surgery.

The follow up last 28 days with 4 visits (D7, D14, D21 and D28).

RESPIMER® NetiFlow® : device of class I, with CE mark, in the indication of sinus postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 65 years of age
* Subject in need of sinus surgery as bilateral total ethmoidectomy using an endoscopic endonasal approach whose pathology is the result of a:

  * Sinonasal polyposis alone
  * Sinonasal polyposis associated with asthma and / or intolerance to NSAIDs
* Free and informed written consent
* Member or beneficiary of a social security program

Exclusion Criteria:

* Oral corticosteroid treatment since less than 2 months
* Premenopausal women not using effective contraception (oral or intrauterine device)
* Pregnant or nursing women
* Uncontrolled diabetes (not treated or stabilized by treatment)
* HIV-positive status
* Autoimmune diseases affecting the nose and/or sinuses, immune dysfunctions (Wegener's granulomatosis, Churg-Strauss syndrome, Common Variable Immunodeficiency, sarcoidosis...), or malignant diseases (unclear histology)
* All contraindication of RESPIMER® NetiFlow®
* All diseases resulting in difficulty coughing or swallowing
* Ongoing or past radiation treatment to the head and neck
* Ongoing or recent chemotherapy (within a three-month period)
* Subjects using anticoagulants
* Subjects taking part in another study that includes an exclusion period coinciding with that of the run-in period of this study
* Subjects placed under judicial protection
* Subjects who suffer from severe physical or psychological problems and whose condition can, according to the investigator, affect compliance with the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Superior healing of nasal mucosa repair 14 days following endoscopic sinus surgery, between the RESPIMER® NetiFlow® solution and the saline solution arms | D14 meaning 14 days (plus or minus 3 days) after surgery
  Based on a ≥8 points difference in the total RHINO QoL score between the two groups.

SECONDARY OUTCOMES:
Efficacy in optimizing airway clearance and restoring respiratory health, as well as overall quality of life | Pre-inclusion, D7, D14, D21 and D28
  Compare the efficacy of RESPIMER® NetiFlow® versus saline solutions in optimizing airway clearance and restoring respiratory health, as well as overall quality of life using:
  * RHINO QoL scores (a self-report of nasal congestion, facial pain, anterior and posterior rhinorrhea).
  * NOSE nasal obstruction scores.
Assess and compare the crusting | Pre-inclusion, D7, D14, D21 and D28
  Assess and compare the crusting with :
  * The number of patients with (whether or not obstruction exists) and without crusting.
  * How many days it takes for the crusting to disappear and/or the difference in the total number of care days
Assess and compare the tolerability | Pre-inclusion, D7, D14, D21 and D28
  Assess and compare the tolerability of RESPIMER® NetiFlow® versus saline solutions using a Visual Analog Scale (VAS) (burning sensation in the nose, alterations in taste and smell and epistaxis) (patient record).
Additional details on duration of nasal washes | D7, D14, D21 and D28 after surgery
  Provide additional details on the duration of nasal washes according to the approved indication (patient record).
Satisfaction and perceived efficacy of the nasal solution | D7, D14, D21 and D28 after surgery
  VAS numerical values assessing the level of patient satisfaction and perceived efficacy in regard to the nasal solution that was used by each group (patient's Case report Form).
Satisfaction, convenience, ease of administration and ease of cleaning of the RESPIMER® NetiFlow® device | D7, D14, D21 and D28 after surgery
  VAS numerical values assessing the RESPIMER® NetiFlow® device in terms of satisfaction, convenience, ease of administration and ease of cleaning (patient's Case report Form).
Assess functionality of nasal lining | D-1, D14, and D21
  Assess functionality of nasal lining by evaluating mucociliary clearance by rhinoscintigraphy for all patients in the 2 Bordeaux centers' (Bordeaux University Hospital and Saint-Augustin Private Hospital):
  * D-1 only for center's Bordeaux, 10 patients in each group (20 patients in total)
  * D14 and D21 for all Bordeaux patients', estimated at 50 patients (15 in each group and in addition the same 10 patients of the D-1 visit, in each group).
Efficacy in improving the trophicity of the nasal mucosa within the operated area | D14, D21 and D28
  Assess the efficacy of RESPIMER® NetiFlow® versus saline solutions in improving the trophicity of the nasal mucosa within the operated area, using a Lund-Kennedy endoscopic score (20 points).

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic LE TAILLANDIER de GABORY, MD, PhD, Principal Investigator — Coordinator Investigator
Locations (8):
- France (8):
  - Service d'Oto-rhino-laryngologie - Clinique Saint-Augustin, Bordeaux, Gironde
  - Service d'Oto-rhino-laryngologie et Chirurgie cervico-faciale - Hôpital Pellegrin, Bordeaux, Gironde
  - ORL et Chirurgie Cervico-faciale - Pôle Voies Respiratoires - CHU Toulouse, Toulouse, Haute-Garonne
  - Service d'ORL et Chirurgie cervico faciale - CHRU Tours, Tours, Indre-et-Loire
  - Service d'oto-rhino-laryngologie - CHU de Nantes, Nantes, Loire-Atlantique
  - Service ORL et Chirurgie Cervico-faciale - CHRU Nancy, Nancy, Meurthe-et-Moselle
  - Service ORL et Chirurgie cervico-faciale - CHRU Lille, Lille, Nord
  - ORL et Chirurgie Cervico-faciale - Centre Hospitalier Intercommunal (CHI) de Créteil, Créteil, Val-de-Marne

REFERENCES:
- [Background] Homer JJ, England RJ, Wilde AD, Harwood GR, Stafford ND. The effect of pH of douching solutions on mucociliary clearance. Clin Otolaryngol Allied Sci. 1999 Aug;24(4):312-5. doi: 10.1046/j.1365-2273.1999.00265.x. PMID 10472466
- [Result] Aarbiou J, Verhoosel RM, Van Wetering S, De Boer WI, Van Krieken JH, Litvinov SV, Rabe KF, Hiemstra PS. Neutrophil defensins enhance lung epithelial wound closure and mucin gene expression in vitro. Am J Respir Cell Mol Biol. 2004 Feb;30(2):193-201. doi: 10.1165/rcmb.2002-0267OC. Epub 2003 Jul 18. PMID 12871849
- [Result] Adam P, Stiffman M, Blake RL Jr. A clinical trial of hypertonic saline nasal spray in subjects with the common cold or rhinosinusitis. Arch Fam Med. 1998 Jan-Feb;7(1):39-43. doi: 10.1001/archfami.7.1.39. PMID 9443697
- [Result] Bardou O, Trinh NT, Brochiero E. Molecular diversity and function of K+ channels in airway and alveolar epithelial cells. Am J Physiol Lung Cell Mol Physiol. 2009 Feb;296(2):L145-55. doi: 10.1152/ajplung.90525.2008. Epub 2008 Dec 5. PMID 19060226
- [Result] Bernstein IL. Is the use of benzalkonium chloride as a preservative for nasal formulations a safety concern? A cautionary note based on compromised mucociliary transport. J Allergy Clin Immunol. 2000 Jan;105(1 Pt 1):39-44. doi: 10.1016/s0091-6749(00)90175-1. PMID 10629450
- [Result] Bieger-Farhan AK, Nichani J, Willatt DJ. Nasal septal mucosal contact points: associated symptoms and sinus CT scan scoring. Clin Otolaryngol Allied Sci. 2004 Apr;29(2):165-8. doi: 10.1111/j.0307-7772.2004.00774.x. PMID 15113304
- [Result] Boek WM, Keles N, Graamans K, Huizing EH. Physiologic and hypertonic saline solutions impair ciliary activity in vitro. Laryngoscope. 1999 Mar;109(3):396-9. doi: 10.1097/00005537-199903000-00010. PMID 10089964
- [Result] Braiman A, Priel Z. Efficient mucociliary transport relies on efficient regulation of ciliary beating. Respir Physiol Neurobiol. 2008 Nov 30;163(1-3):202-7. doi: 10.1016/j.resp.2008.05.010. Epub 2008 May 22. PMID 18586580
- [Result] Britton J, Pavord I, Richards K, Wisniewski A, Knox A, Lewis S, Tattersfield A, Weiss S. Dietary magnesium, lung function, wheezing, and airway hyperreactivity in a random adult population sample. Lancet. 1994 Aug 6;344(8919):357-62. doi: 10.1016/s0140-6736(94)91399-4. PMID 7914305
- [Result] Buchanan PJ, McNally P, Harvey BJ, Urbach V. Lipoxin A(4)-mediated KATP potassium channel activation results in cystic fibrosis airway epithelial repair. Am J Physiol Lung Cell Mol Physiol. 2013 Jul 15;305(2):L193-201. doi: 10.1152/ajplung.00058.2013. Epub 2013 May 17. PMID 23686859
- [Result] Burgel PR, Nadel JA. Roles of epidermal growth factor receptor activation in epithelial cell repair and mucin production in airway epithelium. Thorax. 2004 Nov;59(11):992-6. doi: 10.1136/thx.2003.018879. PMID 15516478
- [Result] Campos J, Heppt W, Weber R. Nasal douches for diseases of the nose and the paranasal sinuses--a comparative in vitro investigation. Eur Arch Otorhinolaryngol. 2013 Nov;270(11):2891-9. doi: 10.1007/s00405-013-2398-z. Epub 2013 Feb 28. PMID 23455580
- [Result] Chen EY, Yang N, Quinton PM, Chin WC. A new role for bicarbonate in mucus formation. Am J Physiol Lung Cell Mol Physiol. 2010 Oct;299(4):L542-9. doi: 10.1152/ajplung.00180.2010. Epub 2010 Aug 6. PMID 20693315
- [Result] Christopher K, Chang J, Goldberg J. Stimulation of cilia beat frequency by serotonin is mediated by a Ca2+ influx in ciliated cells of Helisoma trivolvis embryos. J Exp Biol. 1996;199(Pt 5):1105-13. doi: 10.1242/jeb.199.5.1105. PMID 9318930
- [Result] Ciarallo L, Sauer AH, Shannon MW. Intravenous magnesium therapy for moderate to severe pediatric asthma: results of a randomized, placebo-controlled trial. J Pediatr. 1996 Dec;129(6):809-14. doi: 10.1016/s0022-3476(96)70023-9. PMID 8969721
- [Result] Clark AB, Randell SH, Nettesheim P, Gray TE, Bagnell B, Ostrowski LE. Regulation of ciliated cell differentiation in cultures of rat tracheal epithelial cells. Am J Respir Cell Mol Biol. 1995 Mar;12(3):329-38. doi: 10.1165/ajrcmb.12.3.7873199.
- [Result] Clarke RW, Jones AS. Nasal airflow sensation. Clin Otolaryngol Allied Sci. 1995 Apr;20(2):97-9. doi: 10.1111/j.1365-2273.1995.tb00022.x. No abstract available. PMID 7634531
- [Result] Coraux C, Hajj R, Lesimple P, Puchelle E. [Repair and regeneration of the airway epithelium]. Med Sci (Paris). 2005 Dec;21(12):1063-9. doi: 10.1051/medsci/200521121063. French. PMID 16324647
- [Result] Coraux C, Martinella-Catusse C, Nawrocki-Raby B, Hajj R, Burlet H, Escotte S, Laplace V, Birembaut P, Puchelle E. Differential expression of matrix metalloproteinases and interleukin-8 during regeneration of human airway epithelium in vivo. J Pathol. 2005 Jun;206(2):160-9. doi: 10.1002/path.1757. PMID 15806599
- [Result] Cordray S, Harjo JB, Miner L. Comparison of intranasal hypertonic dead sea saline spray and intranasal aqueous triamcinolone spray in seasonal allergic rhinitis. Ear Nose Throat J. 2005 Jul;84(7):426-30. PMID 16813032
- [Result] Di Benedetto G, Magnus CJ, Gray PT, Mehta A. Calcium regulation of ciliary beat frequency in human respiratory epithelium in vitro. J Physiol. 1991 Aug;439:103-13. doi: 10.1113/jphysiol.1991.sp018659. PMID 1895234
- [Result] Dorscheid DR, Wojcik KR, Yule K, White SR. Role of cell surface glycosylation in mediating repair of human airway epithelial cell monolayers. Am J Physiol Lung Cell Mol Physiol. 2001 Oct;281(4):L982-92. doi: 10.1152/ajplung.2001.281.4.L982. PMID 11557602
- [Result] Dupuit F, Gaillard D, Hinnrasky J, Mongodin E, de Bentzmann S, Copreni E, Puchelle E. Differentiated and functional human airway epithelium regeneration in tracheal xenografts. Am J Physiol Lung Cell Mol Physiol. 2000 Jan;278(1):L165-76. doi: 10.1152/ajplung.2000.278.1.L165. PMID 10645904
- [Result] Dwyer TM, Farley JM. Mucus glycoconjugate secretion in cool and hypertonic solutions. Am J Physiol. 1997 Jun;272(6 Pt 1):L1121-5. doi: 10.1152/ajplung.1997.272.6.L1121. PMID 9227513
- [Result] England RJ, Anthony R, Homer JJ, Martin-Hirsch DP. Nasal pH and saccharin clearance are unrelated in the physiologically normal nose. Rhinology. 2000 Jun;38(2):66-7. PMID 10953843
- [Result] Evans MJ, Cox RA, Shami SG, Wilson B, Plopper CG. The role of basal cells in attachment of columnar cells to the basal lamina of the trachea. Am J Respir Cell Mol Biol. 1989 Dec;1(6):463-9. doi: 10.1165/ajrcmb/1.6.463. PMID 2637758
- [Result] Evans MJ, Cox RA, Burke AS, Moller PC. Differentiation of anchoring junctions in tracheal basal cells in the growing rat. Am J Respir Cell Mol Biol. 1992 Feb;6(2):153-7. doi: 10.1165/ajrcmb/6.2.153. PMID 1540378
- [Result] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Result] Freeman SR, Sivayoham ES, Jepson K, de Carpentier J. A preliminary randomised controlled trial evaluating the efficacy of saline douching following endoscopic sinus surgery. Clin Otolaryngol. 2008 Oct;33(5):462-5. doi: 10.1111/j.1749-4486.2008.01806.x. PMID 18983380
- [Result] Friedman M, Vidyasagar R, Joseph N. A randomized, prospective, double-blind study on the efficacy of dead sea salt nasal irrigations. Laryngoscope. 2006 Jun;116(6):878-82. doi: 10.1097/01.mlg.0000216798.10007.76. PMID 16735920
- [Result] Friedman M, Hamilton C, Samuelson CG, Maley A, Wilson MN, Venkatesan TK, Joseph NJ. Dead Sea salt irrigations vs saline irrigations with nasal steroids for symptomatic treatment of chronic rhinosinusitis: a randomized, prospective double-blind study. Int Forum Allergy Rhinol. 2012 May-Jun;2(3):252-7. doi: 10.1002/alr.21003. Epub 2012 Feb 15. PMID 22337474
- [Result] Georgitis JW. Nasal hyperthermia and simple irrigation for perennial rhinitis. Changes in inflammatory mediators. Chest. 1994 Nov;106(5):1487-92. doi: 10.1378/chest.106.5.1487. PMID 7956408
- [Result] Greiff L, Andersson M, Wollmer P, Persson CG. Hypertonic saline increases secretory and exudative responsiveness of human nasal airway in vivo. Eur Respir J. 2003 Feb;21(2):308-12. doi: 10.1183/09031936.03.00290303. PMID 12608446
- [Result] Greiner J, Diezel W. [Inflammation-inhibiting effect of magnesium ions in contact eczema reactions]. Hautarzt. 1990 Nov;41(11):602-5. German. PMID 2276913
- [Result] Harari M, Barzillai R, Shani J. Magnesium in the management of asthma: critical review of acute and chronic treatments, and Deutsches Medizinisches Zentrum's (DMZ's) clinical experience at the Dead Sea. J Asthma. 1998;35(7):525-36. doi: 10.3109/02770909809048955. PMID 9777879
- [Result] Harvey R, Hannan SA, Badia L, Scadding G. Nasal saline irrigations for the symptoms of chronic rhinosinusitis. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD006394. doi: 10.1002/14651858.CD006394.pub2. PMID 17636843
- [Result] Harvey RJ, Goddard JC, Wise SK, Schlosser RJ. Effects of endoscopic sinus surgery and delivery device on cadaver sinus irrigation. Otolaryngol Head Neck Surg. 2008 Jul;139(1):137-42. doi: 10.1016/j.otohns.2008.04.020. PMID 18585576
- [Result] Hofmann T, Gugatschga M, Koidl B, Wolf G. Influence of preservatives and topical steroids on ciliary beat frequency in vitro. Arch Otolaryngol Head Neck Surg. 2004 Apr;130(4):440-5. doi: 10.1001/archotol.130.4.440. PMID 15096427
- [Result] Hogman M, Mork AC, Roomans GM. Hypertonic saline increases tight junction permeability in airway epithelium. Eur Respir J. 2002 Dec;20(6):1444-8. doi: 10.1183/09031936.02.00017202. PMID 12503702
- [Result] Holgate ST. Epithelial damage and response. Clin Exp Allergy. 2000 Jun;30 Suppl 1:37-41. doi: 10.1046/j.1365-2222.2000.00095.x. PMID 10849473
- [Result] Homer JJ, Dowley AC, Condon L, El-Jassar P, Sood S. The effect of hypertonicity on nasal mucociliary clearance. Clin Otolaryngol Allied Sci. 2000 Dec;25(6):558-60. doi: 10.1046/j.1365-2273.2000.00420.x. PMID 11122299
- [Result] Keerl R, Weber R, Muller C, Schick B. [Effectiveness and tolerance of nasal irrigation following paranasal sinus surgery]. Laryngorhinootologie. 1997 Mar;76(3):137-41. doi: 10.1055/s-2007-997402. German. PMID 9213401
- [Result] Keojampa BK, Nguyen MH, Ryan MW. Effects of buffered saline solution on nasal mucociliary clearance and nasal airway patency. Otolaryngol Head Neck Surg. 2004 Nov;131(5):679-82. doi: 10.1016/j.otohns.2004.05.026. PMID 15523448
- [Result] Konig P, Krain B, Krasteva G, Kummer W. Serotonin increases cilia-driven particle transport via an acetylcholine-independent pathway in the mouse trachea. PLoS One. 2009;4(3):e4938. doi: 10.1371/journal.pone.0004938. Epub 2009 Mar 17. PMID 19290057
- [Result] Krayenbuhl M, Seppey M. [Efficacy of Rhinomer Force 3 in the postoperative course of endonasal surgery]. Rev Med Suisse Romande. 1995 Mar;115(3):249-52. No abstract available. French. PMID 7777766
- [Result] Lackie PM, Baker JE, Gunthert U, Holgate ST. Expression of CD44 isoforms is increased in the airway epithelium of asthmatic subjects. Am J Respir Cell Mol Biol. 1997 Jan;16(1):14-22. doi: 10.1165/ajrcmb.16.1.8998074.
- [Result] Laoukili J, Perret E, Willems T, Minty A, Parthoens E, Houcine O, Coste A, Jorissen M, Marano F, Caput D, Tournier F. IL-13 alters mucociliary differentiation and ciliary beating of human respiratory epithelial cells. J Clin Invest. 2001 Dec;108(12):1817-24. doi: 10.1172/JCI13557. PMID 11748265
- [Result] Larbi KY, Gomperts BD. Complex pattern of inhibition by Mg2+ of exocytosis from permeabilised eosinophils. Cell Calcium. 1997 Mar;21(3):213-9. doi: 10.1016/s0143-4160(97)90045-2. PMID 9105730
- [Result] Lee MK, Yoo JW, Lin H, Kim YS, Kim DD, Choi YM, Park SK, Lee CH, Roh HJ. Air-liquid interface culture of serially passaged human nasal epithelial cell monolayer for in vitro drug transport studies. Drug Deliv. 2005 Sep-Oct;12(5):305-11. doi: 10.1080/10717540500177009. PMID 16188730
- [Result] Levin R, Braiman A, Priel Z. Protein kinase C induced calcium influx and sustained enhancement of ciliary beating by extracellular ATP. Cell Calcium. 1997 Feb;21(2):103-13. doi: 10.1016/s0143-4160(97)90034-8. PMID 9132293
- [Result] Lee RJ, Harlow JM, Limberis MP, Wilson JM, Foskett JK. HCO3(-) secretion by murine nasal submucosal gland serous acinar cells during Ca2+-stimulated fluid secretion. J Gen Physiol. 2008 Jul;132(1):161-83. doi: 10.1085/jgp.200810017. PMID 18591422
- [Result] Lee JM, Nayak JV, Doghramji LL, Welch KC, Chiu AG. Assessing the risk of irrigation bottle and fluid contamination after endoscopic sinus surgery. Am J Rhinol Allergy. 2010 May-Jun;24(3):197-9. doi: 10.2500/ajra.2010.24.3481. PMID 20537286
- [Result] Lock JY, Wyatt E, Upadhyayula S, Whall A, Nunez V, Vullev VI, Liu H. Degradation and antibacterial properties of magnesium alloys in artificial urine for potential resorbable ureteral stent applications. J Biomed Mater Res A. 2014 Mar;102(3):781-92. doi: 10.1002/jbm.a.34741. Epub 2013 Jun 4. PMID 23564415
- [Result] Luk CK, Dulfano MJ. Effect of pH, viscosity and ionic-strength changes on ciliary beating frequency of human bronchial explants. Clin Sci (Lond). 1983 Apr;64(4):449-51. doi: 10.1042/cs0640449. PMID 6825413
- [Result] Ludwig P, Petrich K, Schewe T, Diezel W. Inhibition of eicosanoid formation in human polymorphonuclear leukocytes by high concentrations of magnesium ions. Biol Chem Hoppe Seyler. 1995 Dec;376(12):739-44. doi: 10.1515/bchm3.1995.376.12.739. PMID 9072050
- [Result] Ma W, Korngreen A, Uzlaner N, Priel Z, Silberberg SD. Extracellular sodium regulates airway ciliary motility by inhibiting a P2X receptor. Nature. 1999 Aug 26;400(6747):894-7. doi: 10.1038/23743. PMID 10476971
- [Result] Mahajan P, Haritos D, Rosenberg N, Thomas R. Comparison of nebulized magnesium sulfate plus albuterol to nebulized albuterol plus saline in children with acute exacerbations of mild to moderate asthma. J Emerg Med. 2004 Jul;27(1):21-5. doi: 10.1016/j.jemermed.2004.02.006. PMID 15219299
- [Result] McDowell EM, Becci PJ, Schurch W, Trump BF. The respiratory epithelium. VII. Epidermoid metaplasia of hamster tracheal epithelium during regeneration following mechanical injury. J Natl Cancer Inst. 1979 Apr;62(4):995-1008. PMID 285300
- [Result] Mickenhagen A, Siefer O, Neugebauer P, Stennert E. [The influence of different alpha-sympathomimetic drugs and benzalkoniumchlorid on the ciliary beat frequency of in vitro cultured human nasal mucosa cells]. Laryngorhinootologie. 2008 Jan;87(1):30-8. doi: 10.1055/s-2007-966891. Epub 2007 Sep 18. German. PMID 17879181
- [Result] Nikolaidis E, Eleftheriadou A, Yiotakis I, Lazaris AC, Agrogianis G, Ferekidou E, Keramaris N, Papalois A, Kandiloros D. Influence of intranasal sterile isotonic sea water applications on xylometazoline administration: an experimental study in pigs. Auris Nasus Larynx. 2010 Feb;37(1):71-6. doi: 10.1016/j.anl.2009.03.006. Epub 2009 May 2. PMID 19414231
- [Result] Olson DE, Rasgon BM, Hilsinger RL Jr. Radiographic comparison of three methods for nasal saline irrigation. Laryngoscope. 2002 Aug;112(8 Pt 1):1394-8. doi: 10.1097/00005537-200208000-00013. PMID 12172251
- [Result] Pigret D, Jankowski R. Management of post-ethmoidectomy crust formation: randomized single-blind clinical trial comparing pressurized seawater versus antiseptic/mucolytic saline. Rhinology. 1996 Mar;34(1):38-40. PMID 8739868
- [Result] Pinto JM, Elwany S, Baroody FM, Naclerio RM. Effects of saline sprays on symptoms after endoscopic sinus surgery. Am J Rhinol. 2006 Mar-Apr;20(2):191-6. PMID 16686387
- [Result] Price D, Bond C, Bouchard J, Costa R, Keenan J, Levy ML, Orru M, Ryan D, Walker S, Watson M. International Primary Care Respiratory Group (IPCRG) Guidelines: management of allergic rhinitis. Prim Care Respir J. 2006 Feb;15(1):58-70. doi: 10.1016/j.pcrj.2005.11.002. Epub 2005 Dec 27. PMID 16701759
- [Result] Proksch E, Nissen HP, Bremgartner M, Urquhart C. Bathing in a magnesium-rich Dead Sea salt solution improves skin barrier function, enhances skin hydration, and reduces inflammation in atopic dry skin. Int J Dermatol. 2005 Feb;44(2):151-7. doi: 10.1111/j.1365-4632.2005.02079.x. PMID 15689218
- [Result] Puddicombe SM, Polosa R, Richter A, Krishna MT, Howarth PH, Holgate ST, Davies DE. Involvement of the epidermal growth factor receptor in epithelial repair in asthma. FASEB J. 2000 Jul;14(10):1362-74. doi: 10.1096/fj.14.10.1362. PMID 10877829
- [Result] Pynnonen MA, Mukerji SS, Kim HM, Adams ME, Terrell JE. Nasal saline for chronic sinonasal symptoms: a randomized controlled trial. Arch Otolaryngol Head Neck Surg. 2007 Nov;133(11):1115-20. doi: 10.1001/archotol.133.11.1115. PMID 18025315
- [Result] Rosenfeld RM. Clinical practice guideline on adult sinusitis. Otolaryngol Head Neck Surg. 2007 Sep;137(3):365-77. doi: 10.1016/j.otohns.2007.07.021. PMID 17765760
- [Result] Rudmik L, Soler ZM, Orlandi RR, Stewart MG, Bhattacharyya N, Kennedy DW, Smith TL. Early postoperative care following endoscopic sinus surgery: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2011 Nov-Dec;1(6):417-30. doi: 10.1002/alr.20072. Epub 2011 Oct 29. PMID 22144050
- [Result] Salib RJ, Talpallikar S, Uppal S, Nair SB. A prospective randomised single-blinded clinical trial comparing the efficacy and tolerability of the nasal douching products Sterimar and Sinus Rinse following functional endoscopic sinus surgery. Clin Otolaryngol. 2013 Aug;38(4):297-305. doi: 10.1111/coa.12132. PMID 23714166
- [Result] Satdhabudha A, Poachanukoon O. Efficacy of buffered hypertonic saline nasal irrigation in children with symptomatic allergic rhinitis: a randomized double-blind study. Int J Pediatr Otorhinolaryngol. 2012 Apr;76(4):583-8. doi: 10.1016/j.ijporl.2012.01.022. Epub 2012 Feb 11. PMID 22326210
- [Result] Scadding GK, Durham SR, Mirakian R, Jones NS, Leech SC, Farooque S, Ryan D, Walker SM, Clark AT, Dixon TA, Jolles SR, Siddique N, Cullinan P, Howarth PH, Nasser SM; British Society for Allergy and Clinical Immunology. BSACI guidelines for the management of allergic and non-allergic rhinitis. Clin Exp Allergy. 2008 Jan;38(1):19-42. doi: 10.1111/j.1365-2222.2007.02888.x. PMID 18081563
- [Result] Schmid A, Salathe M. Ciliary beat co-ordination by calcium. Biol Cell. 2011 Apr;103(4):159-69. doi: 10.1042/BC20100120. PMID 21401526
- [Result] Schumacher S, Roth I, Stahl J, Baumer W, Kietzmann M. Biodegradation of metallic magnesium elicits an inflammatory response in primary nasal epithelial cells. Acta Biomater. 2014 Feb;10(2):996-1004. doi: 10.1016/j.actbio.2013.10.030. Epub 2013 Nov 5. PMID 24211732
- [Result] Seppey M, Schweri T, Hausler R. Comparative randomised clinical study of tolerability and efficacy of Rhinomer Force 3 versus a reference product in post-operative care of the nasal fossae after endonasal surgery. ORL J Otorhinolaryngol Relat Spec. 1996 Mar-Apr;58(2):87-92. doi: 10.1159/000276805. PMID 8736053
- [Result] Shani J, Barak S, Levi D, Ram M, Schachner ER, Schlesinger T, Robberecht H, Van Grieken R, Avrach WW. Skin penetration of minerals in psoriatics and guinea-pigs bathing in hypertonic salt solutions. Pharmacol Res Commun. 1985 Jun;17(6):501-12. doi: 10.1016/0031-6989(85)90123-7. PMID 4023031
- [Result] Slapak I, Skoupa J, Strnad P, Hornik P. Efficacy of isotonic nasal wash (seawater) in the treatment and prevention of rhinitis in children. Arch Otolaryngol Head Neck Surg. 2008 Jan;134(1):67-74. doi: 10.1001/archoto.2007.19. PMID 18209140
- [Result] Subiza JL, Subiza J, Barjau MC, Rodriguez R, Gavilan MJ. Inhibition of the seasonal IgE increase to Dactylis glomerata by daily sodium chloride nasal-sinus irrigation during the grass pollen season. J Allergy Clin Immunol. 1999 Sep;104(3 Pt 1):711-2. doi: 10.1016/s0091-6749(99)70351-9. No abstract available. PMID 10482855
- [Result] Suslu N, Bajin MD, Suslu AE, Ogretmenoglu O. Effects of buffered 2.3%, buffered 0.9%, and non-buffered 0.9% irrigation solutions on nasal mucosa after septoplasty. Eur Arch Otorhinolaryngol. 2009 May;266(5):685-9. doi: 10.1007/s00405-008-0807-5. Epub 2008 Sep 18. PMID 18802718
- [Result] Tabary O, Muselet C, Yvin JC, Halley-Vanhove B, Puchelle E, Jacquot J. Physiomer reduces the chemokine interleukin-8 production by activated human respiratory epithelial cells. Eur Respir J. 2001 Oct;18(4):661-6. doi: 10.1183/09031936.01.00075201. PMID 11716171
- [Result] Tabary O, Muselet C, Miesch MC, Yvin JC, Clement A, Jacquot J. Reduction of chemokine IL-8 and RANTES expression in human bronchial epithelial cells by a sea-water derived saline through inhibited nuclear factor-kappaB activation. Biochem Biophys Res Commun. 2003 Sep 19;309(2):310-6. doi: 10.1016/j.bbrc.2003.07.006. PMID 12951051
- [Result] Talbot AR, Herr TM, Parsons DS. Mucociliary clearance and buffered hypertonic saline solution. Laryngoscope. 1997 Apr;107(4):500-3. doi: 10.1097/00005537-199704000-00013. PMID 9111380
- [Result] Tesfaigzi Y. Roles of apoptosis in airway epithelia. Am J Respir Cell Mol Biol. 2006 May;34(5):537-47. doi: 10.1165/rcmb.2006-0014OC. Epub 2006 Jan 26. PMID 16439804
- [Result] Traissac L, Ohayon-Courtes C, Dufour P, Bordenave L. [Nasal washing with Physiomer ... 10 years later: 1988-1998]. Rev Laryngol Otol Rhinol (Bord). 1999;120(2):133-5. French. PMID 10444989
- [Result] Trinh NT, Prive A, Kheir L, Bourret JC, Hijazi T, Amraei MG, Noel J, Brochiero E. Involvement of KATP and KvLQT1 K+ channels in EGF-stimulated alveolar epithelial cell repair processes. Am J Physiol Lung Cell Mol Physiol. 2007 Oct;293(4):L870-82. doi: 10.1152/ajplung.00362.2006. Epub 2007 Jul 13. PMID 17631610
- [Result] Trinh NT, Prive A, Maille E, Noel J, Brochiero E. EGF and K+ channel activity control normal and cystic fibrosis bronchial epithelia repair. Am J Physiol Lung Cell Mol Physiol. 2008 Nov;295(5):L866-80. doi: 10.1152/ajplung.90224.2008. Epub 2008 Aug 29. PMID 18757521
- [Result] Unal M, Seymen HO. Effect of Ringer-Lactate and isotonic saline solutions on mucociliary clearance of tracheal epithelium: an experimental study in rats. J Laryngol Otol. 2002 Jul;116(7):536-8. doi: 10.1258/002221502760132412. PMID 12238674
- [Result] van de Donk HJ, Zuidema J, Merkus FW. The influence of the pH and osmotic pressure upon tracheal ciliary beat frequency as determined with a new photo-electric registration device. Rhinology. 1980 Jun;18(2):93-104. PMID 7403788
- [Result] Watelet JB, Demetter P, Claeys C, Cauwenberge P, Cuvelier C, Bachert C. Wound healing after paranasal sinus surgery: neutrophilic inflammation influences the outcome. Histopathology. 2006 Jan;48(2):174-81. doi: 10.1111/j.1365-2559.2005.02310.x. PMID 16405666
- [Result] Wei CC, Adappa ND, Cohen NA. Use of topical nasal therapies in the management of chronic rhinosinusitis. Laryngoscope. 2013 Oct;123(10):2347-59. doi: 10.1002/lary.24066. Epub 2013 Apr 1. PMID 23553558
- [Result] Wormald PJ, Cain T, Oates L, Hawke L, Wong I. A comparative study of three methods of nasal irrigation. Laryngoscope. 2004 Dec;114(12):2224-7. doi: 10.1097/01.mlg.0000149463.95950.c5. PMID 15564850
- [Result] Yeh TH, Tsai CH, Chen YS, Hsu WC, Cheng CH, Hsu CJ, Lee SY. Increased communication among nasal epithelial cells in air-liquid interface culture. Laryngoscope. 2007 Aug;117(8):1439-44. doi: 10.1097/MLG.0b013e318063e84f. PMID 17572641
- [Result] Zahm JM, Kaplan H, Herard AL, Doriot F, Pierrot D, Somelette P, Puchelle E. Cell migration and proliferation during the in vitro wound repair of the respiratory epithelium. Cell Motil Cytoskeleton. 1997;37(1):33-43. doi: 10.1002/(SICI)1097-0169(1997)37:13.0.CO;2-I. PMID 9142437
- [Result] Zsembery A, Boyce AT, Liang L, Peti-Peterdi J, Bell PD, Schwiebert EM. Sustained calcium entry through P2X nucleotide receptor channels in human airway epithelial cells. J Biol Chem. 2003 Apr 11;278(15):13398-408. doi: 10.1074/jbc.M212277200. Epub 2003 Feb 3. PMID 12566439
- [Result] Zsembery A, Fortenberry JA, Liang L, Bebok Z, Tucker TA, Boyce AT, Braunstein GM, Welty E, Bell PD, Sorscher EJ, Clancy JP, Schwiebert EM. Extracellular zinc and ATP restore chloride secretion across cystic fibrosis airway epithelia by triggering calcium entry. J Biol Chem. 2004 Mar 12;279(11):10720-9. doi: 10.1074/jbc.M313391200. Epub 2003 Dec 29. PMID 14701827